CLINICAL TRIAL: NCT05132946
Title: Ultrasound-guided Erector Spinae Plane Block: A Comparative Study to Assess Its Analgesic Efficacy in Pediatric Patients Undergoing Aortic Coarctation Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, samar mohammed, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAMSU R 167/2021
Record Dates: First submitted 2021-11-01; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (B): will receive erector spinae plane block. (Active Comparator): unilateral ultrasound-guided erector spinae plane block using bupivacaine 0.25% (on the left side) with total volume 0.5 ml/kg and a maximum dose of 2 mg/kg of bupivacaine in erector spinae plane block group patients
  Interventions: Procedure: Nerve block
- • Group (C): will not receive any block. (No Intervention)

INTERVENTIONS:
Procedure: Nerve block — unilateral ultrasound-guided erector spinae plane block using bupivacaine 0.25% (on the left side) with total volume 0.5 ml/kg and a maximum dose of 2 mg/kg of bupivacaine in erector spinae plane block group patients
  Arms: Group (B): will receive erector spinae plane block.

SUMMARY:
The study will include 40 patients who fulfil all the points in the inclusion and exclusion criteria will be randomized into two equal groups, each consisting of 20 patients, namely group (B) and group (C).

* Group (B): will receive erector spinae plane block.
* Group (C): will not receive any block. Postoperative pain score will be assessed using the FLACC scale or Face, Legs, Activity, Cry, Consolability scale immediately after extubation and at 1, 2, 4, 6, 8, 12, 18, and 24 hours. Routine postoperative analgesia in the form of intravenous paracetamol 7.5 mg/kg/6 hours will be given to all patients (the first dose is given after skin closure). Rescue analgesia in the form of 1 ug/kg fentanyl intravenously for patients if FLACC scale > 4, and the time for the first rescue analgesic administration will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients presented for aortic coarctation repair via left thoracotomy.

Exclusion Criteria:

Hypersensitivity to local anesthetic.

* Mental or neurologic disorders.
* Preoperative critically ill patients.
* Parents or legal guardian refusal.
* Infection at the site of injection.
* Any liver disease.
* Any coagulopathy.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-10 (Estimated)

PRIMARY OUTCOMES:
The number of times for usage of fentanyl in postoperative period | in the first 12 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Soliman, Cairo, Nasr City, Egypt